CLINICAL TRIAL: NCT00235599
Title: The Insulin-Like Growth Factor Binding Protein-3 Test: A New Tool for the Diagnosis of Growth Hormone Deficiency in Children.
Brief Title: The IGFBP-3 Stimulation Test: A New Tool for the Diagnosis of Growth Hormone Deficiency in Children.
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Other Study IDs: 305-SG01; H-11757
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Short Stature; Growth Hormone Deficiency
Keywords: Growth; Hormone; Deficiency
MeSH Terms: conditions — Dwarfism; Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: IGFBP-3 Stimulation Test

SUMMARY:
This project is designed to answer the question: Is there an acute IGFBP-3 response in normal children?

Our specific hypothesis states that under the influence of growth hormone secretagogues, intact IGFBP-3 molecule will undergo proteolysis and liberate IGFBP-3 fragments, along with other components of the ternary complex. This proteolysis will result in measurable rise in IGFBP-3, which will indicate the subject's growth hormone status. Short children with growth hormone deficiency will not show an IGFBP-3 response.

DETAILED DESCRIPTION:
The diagnosis of growth hormone deficiency is problematic, given the shortcoming of the standard growth hormone stimulation test. This study is designed to investigate a new tool for the diagnosis of growth hormone deficiency.

Ten short, prepubertal children, who fulfill the inclusion criteria, will undergo a two-secretagogue standard growth hormone stimulation test, and an insulin like growth factor binding protein-3 (IGFBP-3) stimulation test simultaneously. During this test, components of the ternary complex moieties, viz, insulin-like growth factor-I (IGF-I), IGFBP-3 and acid labile subunit (ALS) will also be measured along with growth hormone.

The aim of this study is to detect an acute rise in IGFBP-3 of >15% from baseline.

The importance of this study is that it inculcates the specificity and improved sensitivity of stimulated IGFBP-3 in the diagnosis of growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Bone age < 10 years female, < 12 years male
* Pubertal status: Girls: Tanner I for breast development. Boys: testicular volume of ≤ 3 cc, as measured by the standardized orchidometer (Prader type). The onset of pubic hair development up to and including Tanner III is allowed in the study.
* Adequate nutrition: body mass index ≥ 25th percentile for gender.

Exclusion Criteria:

* Syndromic short stature
* Chronic illnesses.
* Other disorders, including osteo- or chondrodystrophies, and endocrine causes of short stature such as Cushing syndrome, and untreated hypothyroidism.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2005-09; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U Nwosu, MD, Principal Investigator — University of Massachusetts, Worcester; Carol A Cicarrelli, RN, Study Director — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Nwosu BU, Soyka LA, Angelescu A, Lee MM. Evidence of insulin-like growth factor binding protein-3 proteolysis during growth hormone stimulation testing. J Pediatr Endocrinol Metab. 2011;24(3-4):163-7. doi: 10.1515/jpem.2011.088. PMID 21648284